CLINICAL TRIAL: NCT01341288
Title: Phase I Study Using EUCLIDIAN Robotic Assistance During Prostate Brachytherapy
Brief Title: Robotic Seed Implantation for Prostate Cancer Brachytherapy
Acronym: EUCLIDIAN
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08F.298; 2007-24 (Other: CCRRC); R01CA091763 (NIH); JT 1232 (Other: JeffTrial Number)
Record Dates: First submitted 2011-03-29; First posted 2011-04-25 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; EUCLIDIAN; Endo-Uro Computed Lattice for Intratumoral Delivery, Implantation, Ablation with Nanosensing; robot; brachytherapy; seed implantation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implant (Experimental): Robotic implantation of brachytherapy seeds to treat prostate cancer
  Interventions: Device: EUCLIDIAN Robot

INTERVENTIONS:
Device: EUCLIDIAN Robot — EUCLIDIAN (Endo-Uro Computed Lattice for Intratumoral Delivery, Implantation, Ablation with Nanosensing) system for placement of radioactive seeds in the prostate
  Other Names: Endo-Uro Computed Lattice for Intratumoral Delivery, Implantation, Ablation with Nanosensing

SUMMARY:
A robotic brachytherapy device will be used to assist physicians in performing seed implantation to the prostate. EUCLIDIAN is the first robotic system designed to allow automatic placement of radioactive seeds by robot and thus reduce operator dependence. The clinical study is designed to evaluate the dosimetric quality, accuracy and patient self-reported quality of life scores after robotic brachytherapy.

DETAILED DESCRIPTION:
EUCLIDIAN (Endo-Uro Computed Lattice for Intratumoral Delivery, Implantation, Ablation with Nanosensing)

The dose-volume histogram parameters of robotic brachytherapy will be compared to historical controls of the study institution. Short-term (<1 yr) health-related quality of life (HRQoL) and changes will be assessed using FACT-P and IPSS self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, adenocarcinoma of the prostate, clinical stage T1c-T2b, NX, N0, M0.
* Zubrod status 0-1.
* Prostate tumor biopsy grading by Gleason score classification is mandatory prior to registration
* No prior pelvic radiation or chemotherapy for any reason; induction hormonal therapy beginning < or = 6 months prior to registration is acceptable.
* Prostate volume < or = 65 cc prior to registration, or planned use of LHRH agonist therapy for reduction of prostate volume. If LHRH agonist therapy is used to reduce prostate volume, then prostate volume must be < or = 65 cc on the routine pre-implant volume study to be eligible for the study.
* Gleason score 6, or Gleason Score 7 if both , or = 33% of biopsy cores contain cancer and PSA level is < or = 10 ng/mL.
* AUA voiding symptoms score < or = 15.
* Prostate specific antigen (PSA) prior to study entry (and prior to any hormone treatment if given); must be < or = 20 ng/ml.
* Patients must sign a study-specific consent form prior to registration (Standard of care: only the standard consent form must be signed).
* Patient must be > or = 40 years old.

Exclusion Criteria:

* Stage T2c, T3 or T4 disease.
* Lymph node involvement (pathological N1)
* Evidence of distant metastases (M1)
* Gleason score 8-10.
* Prostate specific antigen (PSA) prior to study entry > 20 ng/mL.
* AUA voiding symptoms score > 15.
* Radical surgery for carcinoma of the prostate.
* Previous hormonal therapy beginning > 6 months prior to registration
* Previous or concurrent cancers other than basal or squamous cell skin cancers unless disease- free for > or = 5 years.
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up and/or completion of HRQoL questionnaires (not a condition for ineligibility in Standard of care).
* Prior TURP
* Hip prosthesis

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07-29 (Actual); Primary Completion 2015-02-26 (Actual); Study Completion 2015-02-27 (Actual)

PRIMARY OUTCOMES:
Coverage of the prostate by the prescribed radiation dose at V100 | Day 0 and Day 30 post-implant
  The principal endpoint is the dose-volume histogram (DVH) measured at V100 (percent volume of the target receiving the intended dose). These values will also be compared retrospectively to those in the conventional group. Improved quality will be demonstrated by increased V100 in the protocol patients.

SECONDARY OUTCOMES:
Coverage of the prostate by the prescribed radiation dose at D90 | 12 months post-treatment
  The secondary endpoint is the dose-volume histogram (DVH) measured at D90 (dose to 90% of the target volume). These values will also be compared retrospectively to those in the conventional group.
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 12 months
  Patient self-reported, health-related, quality of life measures using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) self-report questionnaire. FACT-P instruments prior to treatment (T0), 1 month (T1), 3 months (T3), 6 months (T6) and 12 months (T12) following treatment with robot-assisted brachytherapy.
International Prostate Symptom Score (IPSS) | 12 months
  Patient self-reported, health-related, quality of life measures using the International Prostate Symptom Score (IPSS) self-report questionnaire. IPSS instruments prior to treatment (T0), 1 month (T1), 3 months (T3), 6 months (T6) and 12 months (T12) following treatment with robot-assisted brachytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Podder TK, Buzurovic I, Huang K, Showalter T, Dicker AP, Yu Y. Reliability of EUCLIDIAN: an autonomous robotic system for image-guided prostate brachytherapy. Med Phys. 2011 Jan;38(1):96-106. doi: 10.1118/1.3523097. PMID 21361179
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org